CLINICAL TRIAL: NCT06861608
Title: A Single-session Intervention Adaptation of the Habit Framework for the Prevention of Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Eating Disorders Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20030734; FP00023118 (Other Grant/Funding Number: National Eating Disorder Association)
Record Dates: First submitted 2025-01-27; First posted 2025-03-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Eating Disorder Not Otherwise Specified
Keywords: prevention of eating disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial to test the acceptability and feasibility of a single-session intervention utilizing the habit framework for adolescents and young adults who are at-risk of developing a restrictive eating disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: psychoeducation experience single-session intervention (SSI) (Experimental): This online randomized controlled trial of a habit training intervention includes one 30-minute session for young adults endorsing high levels of eating pathology. The intervention will occur at one timepoint.
  Interventions: Behavioral: Screening Questionnaire; Behavioral: Pre-Intervention Questionnaires (~10 minutes); Behavioral: SSI (Single-session intervention (~30 minutes) Active arm; Behavioral: End-of-Intervention Questionnaires (~5 minutes)
- Control: will be matched to the SSI by including both reading and writing exercises. (Placebo Comparator): The control intervention will consist of supportive therapy focusing on sharing emotions and include an introduction to emotions, writing about emotions, testimonials from other adolescents about the power of sharing emotions, and an exercise asking adolescents how different situations might make them feel.
  Interventions: Behavioral: Screening Questionnaire; Behavioral: Pre-Intervention Questionnaires (~10 minutes); Behavioral: SSI (Single-session intervention (~30 minutes) control arm; Behavioral: End-of-Intervention Questionnaires (~5 minutes)

INTERVENTIONS:
Behavioral: Screening Questionnaire — Individuals will complete an online screening survey through an online study advertisement to determine initial eligibility. The screening survey will ask participants to report their gender and age and complete the Eating Attitudes Test - 26-item (EAT-26). EAT-26 scores equal to or greater than 20 indicate risk for an eating disorder. EAT-26, participants will meet the "referral criteria" which includes a score of 20 or more or meeting frequency criteria on bingeing, purging, laxative/diuretic use, and/or exercise. If an interested individual is not eligible, they will be notified that they are not currently eligible for the study and provided with resources.
Behavioral: Pre-Intervention Questionnaires (~10 minutes) — Eligible participants will complete pre-intervention questionnaires including demographics and symptom measures.
Behavioral: SSI (Single-session intervention (~30 minutes) Active arm — The SSI will consist of four components: 1)psychoeducation, 2) real-life examples, 3) common questions and misconceptions, and 4) providing advice to other young adults. Psychoeducation will focus on the brain bases of habit formation and EDs, as per REACH+ treatment manual. Participants will then be asked to think of a real-life example of an eating habit in which they have been engaged, such as limiting their intake of dessert foods. Participants will then be provided with REACH+ developed psychoeducation regarding changing habits, including information on competing responses, stimulus control, and exposure. Participants will have the opportunity to write out how they could use one of these strategies to tackle the habit that they previously wrote about. They will be provided with a worksheet to help them move through each aspect of changing their habit based on what they learned.
  Arms: Experimental: psychoeducation experience single-session intervention (SSI)
Behavioral: SSI (Single-session intervention (~30 minutes) control arm — The control condition will be matched to the SSI by including both reading and writing exercises. The control intervention will consist of supportive therapy focusing on sharing emotions and include an introduction to emotions, writing about emotions, testimonials from other adolescents about the power of sharing emotions, and an exercise asking adolescents how different situations might make them feel.
  Arms: Control: will be matched to the SSI by including both reading and writing exercises.
Behavioral: End-of-Intervention Questionnaires (~5 minutes) — Participants will complete additional questionnaires at the end of the intervention, including acceptability ratings and program feedback. Participants will provide an email address at the end of the questionnaires for receipt of four-week follow-up questionnaires.

SUMMARY:
The purpose of this proposal is to launch the first trial of a single-session intervention (SSI) specifically for the prevention of eating disorders (EDs).

DETAILED DESCRIPTION:
The emergence of EDs is bimodal such that there is a period of risk in early adolescence and a period of risk in late adolescence/early adulthood. EDs can lead to significant mental and physical health consequences and have one of the highest mortality rates of any mental illness. Prevention and treatment programs for EDs are fraught with barriers to access, particularly related to seeking care in-person. SSIs have been identified as a pathway to address the gap in care for EDs after showing promise for other psychiatric problems, including depression, anxiety, and suicidality .

ELIGIBILITY:
Inclusion Criteria:

* EAT-26 score ≥ 20 ( EAT-26, participants will meet the "referral criteria" which includes a score of 20 or more or meeting frequency criteria on bingeing, purging, laxative/diuretic use, and/or exercise.)
* English-language fluency, self-reported3
* Access to a phone, tablet, or computer

Exclusion Criteria:

* Failure to correctly complete one of the attention checks in the survey prior to the intervention
* Failure to correctly complete both anagram tasks in the survey prior to the intervention
* Completion of the screening survey or pre-intervention surveys in an improbably fast time

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Eating Attitudes Test - 26-item | Baseline though study completion and up to one month follow-up
  This 26-item measure will be used to assess eating disorder, including bingeing, purging, and exercise behaviors. According to this methodology, individuals who score 20 or more on the test should be interviewed by a qualified professional to determine if they meet the diagnostic criteria for an eating disorder. If you have a low score on the EAT-26 (below 20), you still could have a serious eating problem, so do not let the results deter you from seeking help. For example, some individuals with Binge Eating Disorder (BED) score low on the EAT-26 but may have a serious eating disorder.
The Brief (Seven-item) Eating Disorder Examination Questionnaire | Baseline though study completion and up to one month follow-up
  This measure will be used to assess eating behaviors over the past month. The seven-item version consists of seven items derived from the original Eating Disorder Examination Questionnaire and assesses for dietary restraint, shape/weight overvaluation, and body dissatisfaction. It consists of three subscales: dietary restraint (items 1, 3 and 4), shape/weight overvaluation (items 22 and 23) and body dissatisfaction (items 25 and 26).
Self-report Habit Index | Baseline though study completion and up to one month follow-up
  The self-report habit index measures habit strength, which is the underlying mechanism being targeted in the current intervention. 7-point Likert scale from "strongly disagree" to "strongly agree." Higher scores indicate a stronger habit, suggesting the behavior is more automatic and less consciously controlled.
State Hope Scale - Agency Subscale | Baseline though study completion and up to one month follow-up
  The 3-item agency subscale of the State Hope Scale measures belief in one's capacity to initiate and sustain actions. Research has shown that high agency is predictive of goal-related activities and utilization of coping skills. Higher scores on the agency subscale generally indicate a stronger sense of personal agency and belief in one's ability to take control and actively pursue goals.
Beck Hopelessness Scale - 4-item Version | Baseline though study completion and up to one month follow-up
  This 4-item measure assesses hopelessness about the future with excellent psychometric properties and good internal consistency. typically calculated by summing up the responses to the four selected items, with a potential range from 0 to 4, where higher scores indicate greater levels of hopelessness.
Barriers to Seeking Treatment. | Baseline though study completion and up to one month follow-up
  Help-seeking barriers will be assessed using this 26-item measure that was created in alignment with results of a systematic review of barriers and facilitators to help-seeking in eating disorders. A high score on a barrier-to-treatment scale suggests that the individual perceives that particular factor as a significant obstacle to seeking professional help.
SSI | Baseline though study completion and up to one month follow-up
  The SSI will consist of four components: 1)psychoeducation, 2) real-life examples, 3) common questions and misconceptions, and 4) providing advice to other young adults based on what participants learned throughout the intervention. Psychoeducation will focus on the brain bases of habit formation and EDs, as per REACH+ treatment manual. Participants will then be asked to think of a real-life example of an eating habit in which they have been engaged, such as limiting their intake of dessert foods. Participants will then be provided with REACH+ developed psychoeducation regarding changing habits, including information on competing responses, stimulus control, and exposure. Participants will have the opportunity to write out how they could use one of these strategies to tackle the habit that they previously wrote about. They will be provided with a worksheet to help them move through through each aspect of changing their habit based on what they learned.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Breiner, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided